CLINICAL TRIAL: NCT00894699
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Clinical Efficacy, Safety and Tolerability of ARX-F03 Sublingual Sufentanil/Triazolam NanoTabs™ in Patients Undergoing an Elective Abdominal Liposuction Procedure
Brief Title: A Study to Evaluate the Clinical Efficacy, Safety and Tolerability of ARX-F03 Sublingual Sufentanil/Triazolam NanoTab™ in Patients Undergoing an Elective Abdominal Liposuction Procedure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARX-C-007
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-05

CONDITIONS: Sedation; Anxiety; Pain
Keywords: procedural sedation
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): single dose of sublingual Sufentanil 15 mcg/Triazolam 200 mcg NanoTab™
  Interventions: Drug: Sublingual Sufentanil/Triazolam NanoTab™ (ARX-F03)
- 2 (Placebo Comparator): single dose of sublingual Placebo NanoTab™
  Interventions: Drug: Placebo NanoTab™

INTERVENTIONS:
Drug: Sublingual Sufentanil/Triazolam NanoTab™ (ARX-F03) — Single dose of sublingual Sufentanil 15 mcg/Triazolam 200 mcg NanoTab™
  Arms: 1
Drug: Placebo NanoTab™ — Single dose of sublingual placebo NanoTab™
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a study medication that contains a combination of a pain medication, sufentanil, and a sedative, triazolam. This drug is being designed to provide mild sedation as well as reduce anxiety and pain before and during a procedure (in this case elective abdominal liposuction).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have provided written informed consent to participate in the study.
2. Male or female patient between 18 to 60 (inclusive) years of age.
3. Patient is planning to undergo an elective outpatient abdominal liposuction procedure.
4. Patient must be classified as American Society of Anesthesiologists (ASA) class I - III.
5. Patient must have Body Mass Index [BMI = weight (kg)/height (m2)] between 20 and 35, inclusively.
6. Female patients of childbearing potential must be using an effective method of birth control at the time of the screening visit and for 30 days following the dosing of study medication. Acceptable methods of birth control include oral or transdermal contraceptives, condom, spermicidal foam, intrauterine device (IUD), progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or postmenopausal for ≥1 year, must be specified. Patients using hormonal forms of contraception must also be willing to use a barrier method of contraception from screening through 30 days following the dose of study medication.
7. Patient is willing to receive antibiotics as per the normal practice of the surgeon.
8. Patient understands that preoperative analgesics or anxiolytics are not permitted.
9. Patient is willing to avoid caffeine and alcohol use within 24 hours before the procedure.
10. The patient must be willing and able to understand the study procedures and the use of pain and anxiety scales, and to communicate meaningfully with the study personnel.
11. The patient must have a caregiver available to escort the patient home following the procedure.

Exclusion Criteria:

1. Patient who is expected to require less than 400 cc or more than 700 cc of abdominal fat removal during the procedure.
2. Patient has previously not responded to opioid analgesics for treatment of pain.
3. Patient has previously not responded to benzodiazepines for treatment of anxiety.
4. Patient is currently taking any opioid or has taken any opioid for more than 7 consecutive days of daily use within the past 3 months prior to the procedure.
5. Patient is currently taking any benzodiazepine or has taken any benzodiazepine for more than 7 consecutive days within the past 3 months prior to the procedure.
6. Patient is taking monoamine oxidase inhibitors (MAOIs), or have taken MAOIs within 14 days prior to enrolling in the study.
7. Patient has an allergy or hypersensitivity to opioids.
8. Patient who is currently taking anti-inflammatory drugs, including steroids.
9. Use of drugs which are P450 3A4 inducers or inhibitors within 30 days of dosing including alprazolam, chlorpheniramine, cimetidine, fluoxetine, haloperidol, ketoconazole, itraconazole, erythromycin, clarithromycin, sildenafil, simvastatin, St. John's Wort.
10. Patient who is taking calcium channel blockers or beta blockers.
11. Patient who will consume grapefruit, or products made with grapefruit, within 3 days of study medication dosing.
12. Patient with a history of chronic obstructive pulmonary disease (COPD) or any other respiratory condition or active pulmonary disease.
13. Patient currently has sleep apnea that has been documented by a sleep laboratory study.
14. Patient is a woman who is pregnant or lactating.
15. Patient has a history of an anxiety disorder.
16. Patients with oral mucositis or stomatitis.
17. Patient has a history of drug, prescription medicine, or alcohol abuse within the past 2 years.
18. Patient used an investigational drug or device within 30 days of screening visit.
19. Patient has undergone a liposuction procedure previously.
20. Patient has a history of migraine or chronic headache.
21. Patient who has a positive urine screen for drugs of abuse at screening or on the day of procedure.
22. Patient who has a positive alcohol screen on the day of the procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Palmer, M.D., PhD, Study Director — Talphera, Inc
Locations (1):
- Lotus Clinical Research, Inc., Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated 22 June 2009 and completed 11 September 2009. One clinical research center participated in the study
Pre-assignment Details: Patients were to be between 18 and 60 years of age, generally healthy, and who are expected to require more than 400 cc or less than 700 cc of abdominal fat removal during the procedure.
Groups:
- Sufentanil 15 mcg/Triazolam 200 mcg NanoTab™: Single dose of sublingual Sufentanil 15 mcg/Triazolam 200 mcg NanoTab™
- Single Dose of Placebo NanoTab™: Single dose of sublingual Placebo NanoTab™
Period: Overall Study
Arm/Group | Sufentanil 15 mcg/Triazolam 200 mcg NanoTab™ | Single Dose of Placebo NanoTab™
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sufentanil/Triazolam NanoTab™: Single dose of sublingual Sufentanil/Triazolam 15/200 mcg NanoTab™
- Placebo: Single dose of Placebo
- Total: Total of all reporting groups
Arm/Group | Sufentanil/Triazolam NanoTab™ | Placebo | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (9.8) | 37.3 (7.7) | 36.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Summed Richmond Agitation Sedation Score (RASS) Over the 4-hour Study Period (SRS-4)
Description: The primary efficacy endpoint of the study is the sedation level as assessed by the 10-point RASS, where unarousable is graded as minus 5 (- 5) and combative is graded as plus 4 (+ 4). The RASS was assessed at 15 time points throughout the four hour study period.
Time Frame: 4 hour study period
Population: ITT population were those patients that took at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Sublingual Sufentanil 15 mcg/Triazolam NanoTab™ 200 mcg: Single dose of sublingual Sufentanil 15 mcg/Triazolam 200 mcg NanoTab™
Arm/Group | Sublingual Sufentanil 15 mcg/Triazolam NanoTab™ 200 mcg | Placebo NanoTab™
Number analyzed (Participants) | 21 | 19
units on a scale | -5.44 (.82) | 0.79 (.86)
Statistical Analysis 1: Comparison: Sublingual Sufentanil 15 mcg/Triazolam NanoTab™ 200 mcg vs Placebo NanoTab™; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Sublingual Sufentanil 15 mcg/Triazolam NanoTab™ 200 mcg vs Placebo NanoTab™; Test type: Superiority or Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: 4 hours.
Description: A telephone call was placed to each patient 24 hours after dosing to inquire about the patients' overall health. If AEs were reported, they were documented in the clinical database.
Groups:
- Sufentanil/Triazolam NanoTab™: Single dose of sublingual Sufentanil 15 mcg/Triazolam 200 mcg NanoTab™
Arm/Group | Sufentanil/Triazolam NanoTab™ | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 5/21 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil/Triazolam NanoTab™ (N=21) | Placebo (N=19)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — All events listed in this table were considered possibly or probably related to study drug
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Hypoxia (Vascular disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other